CLINICAL TRIAL: NCT00037999
Title: The Effect of Testosterone Supplementation on Rehabilitation Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E2419R
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-05

CONDITIONS: Aging; Frail Elderly; Rehabilitation
Keywords: Muscle strength; Testosterone; Rehabilitation; Impaired muscle strength

INTERVENTIONS:
Procedure: Testosterone supplement

SUMMARY:
The objective of this project is to determine the safety and efficacy of testosterone supplementation as an adjunct to traditional rehabilitation therapy in the care of deconditioned older men. Our long range goal is to determine whether other hormones (e.g., combined testosterone and growth hormone) are helpful as an adjunct to traditional rehabilitation therapy.

This project is important to the VA health care system because 38% of American veterans are aged (age > 65 years), bioavailable testosterone is diminished in older age men, low testosterone is associated with impaired muscle strength, and lack of muscle strength hinders rehabilitation. Older men who are not successfully rehabilitated often get admitted to nursing homes for long term care, at a cost of approximately $40,000/year. Payment for long term care is currently one of our most difficult health care problems. If testosterone supplementation improves rehabilitation outcomes, as our pilot data suggest it will, patients will be more satisfied and long-term care financial resources will be saved.

We will conduct a randomized, placebo-controlled trial to test the hypothesis that supplementation with testosterone improves rehabilitation outcomes in deconditioned older men. Specifically, we will screen all hospitalized older men with delayed discharge from the hospital (> 7 day hospital stay). Men who have at least one new impairment in their ability to perform activities of daily living (e.g., inability to walk), low serum testosterone concentration, and no contraindications (e.g., prostate or breast cancer) will be offered the opportunity to participate. Study participants will be randomized to receive either testosterone (5 mg transdermally each night) or placebo (matching transdermal patch) daily in a double-blind fashion for the duration of their hospital course (expected average duration of study is 29 days). Subjects will then receive their rehabilitation as usual, with all members of the health care team blinded as to whether the subject is receiving testosterone or placebo. At baseline, weekly, at discharge, and at 6 and 12 months after discharge, subjects will be assessed using validated measures (i.e., Functional Independence Measure - FIM). Our hypothesis is that testosterone supplementation, as an adjunct to traditional rehabilitation therapy, will improve rehabilitation outcomes.

DETAILED DESCRIPTION:
Our overall goal is to determine the safety and efficacy of testosterone supplementation as an adjunct to traditional rehabilitation therapy on health outcomes in deconditioned older men. Specifically, we will conduct a randomized, placebo-controlled trial to test the hypothesis that supplementation with testosterone improves rehabilitation outcomes in deconditioned older men. We will use objective validated measures (i.e., FIM, muscle strength) to assess health outcomes.

We will begin enrolling subjects within three months of receipt of funding, and study 60 subjects (30 in each group) within 24 months. All subjects will undergo follow-up evaluation 6 and 12 months after completion of inpatient rehabilitation and cessation of testosterone supplementation. Therefore, this project will be completed within 3 years. Our short term goal (within 3 years) is to delineate the safety and efficacy of testosterone supplementation on rehabilitation outcomes in deconditioned older men. Our long range goal is to determine whether other hormones (e.g., combined testosterone and growth hormone) are helpful as an adjunct to traditional rehabilitation therapy in the care of older men

ELIGIBILITY:
Older men with diminished muscle strength

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-04; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D. Special Assistant to the Director — Program Analysis and review Section (PARS), VA Rehabilitation Research & Development Service; Vicki Mongiardo, Program Analyst — Program Analysis and Review Section (PARS), VA Rehabilitation Research and Development Service
Locations (1):
- VA Medical Center, Richmond, Virginia, United States